CLINICAL TRIAL: NCT01217125
Title: CLINICAL TRIAL TO DETERMINE THE EFFICACY AND SAFETY OF RAPAMYCIN IN ANGIOMYOLIPOMAS IN PATIENTS WITH TUBEROUS SCLEROSIS
Brief Title: Rapamycin In Angiomyolipomas In Patients With Tuberous Sclerosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundacio Puigvert (Other)
Collaborators: Ministry of Health, Spain (Other Government)
Responsible Party: Principal Investigator, Roser Torra, MD, PhD, Fundacio Puigvert
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT 2007-005978-30
Record Dates: First submitted 2010-10-06; First posted 2010-10-08 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: Angiomyolipoma
Keywords: tuberousclerosis, angiomyolipoma, rapamycin
MeSH Terms: conditions — Angiomyolipoma | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Sirolimus — plasma levels between 4 and 8
  Other Names: Rapamune

SUMMARY:
The purpose of this study is to determine whether rapamycin is safe and effective in the treatment of renal angiomyolipomas in patients with tuberousclerosis.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of tuberousclerosis Angiomyolipoma >2cm age>10 years

Exclusion Criteria:

Creatinine >4 No recent AML bleeding No hepatic abnormalities (liver tests 2fold) Hematocrit<27% Thrombocytopenia (<100.000/mm3) Leukopenia (<3000/mm3) Ischemic cardiopathy Recent surgery (2 months prior to enrollment) Pregnancy Serum cholesterol over 7.8 mmol/l or hypertriglyceridemia fasten(>4.6 mmol/l) non controlled with drugs malignancy in the previous 2 years allergy to macrolides

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-10; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Angiomyolipoma volume | 2 years
  Measured by MRI

SECONDARY OUTCOMES:
skin lesions, AML complications, | 2 years
  Evaluate skin lesions Collect event realted to AML

CONTACTS AND LOCATIONS:
Overall Officials: Roser Torra, MD,PhD, Principal Investigator — Fundacio Puigvert, Barcelona

REFERENCES:
- [Derived] Cabrera-Lopez C, Marti T, Catala V, Torres F, Mateu S, Ballarin J, Torra R. Assessing the effectiveness of rapamycin on angiomyolipoma in tuberous sclerosis: a two years trial. Orphanet J Rare Dis. 2012 Nov 11;7:87. doi: 10.1186/1750-1172-7-87. PMID 23140536